CLINICAL TRIAL: NCT03207178
Title: Sequential Infusion of Anti-CD19 and Anti-CD20 Chimeric Antigen Receptor(CAR) T Cells Against Relapsed and Refractory B-cell Lymphoma
Brief Title: Sequential Infusion of Anti-CD19 and Anti-CD20 CAR-T Cells Against Relapsed and Refractory B-cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Longyao Biotechnology Inc., Ltd. (Other)
Collaborators: Xuzhou Medical University (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LYCT-1701
Record Dates: First submitted 2017-06-23; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Recurrent or Refractory B Cell Malignancy
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mixed CD19/CD20 CAR-T Transfer (Experimental): Subjects with CD19+/CD20+ B-cell lymphomas will be infused with CD19-targeting CAR T Cells and CD20-targeting CAR T Cells in one time or in parts
  Interventions: Biological: Mixed CD19/CD20 CAR-T Transfer

INTERVENTIONS:
Biological: Mixed CD19/CD20 CAR-T Transfer — Autologous CD19 CAR-T cells and CD20 CAR-T cells with average 1-5*10^6 cells/kg body weight,separately.

SUMMARY:
Cluster of differentiation antigen 19(CD19) specifically presents in B lymphocyte cell lines steadily,while not in most normal tissue,including pluripotent hematopoietic stem cells.Cluster of differentiation antigen 20(CD20) presents in 90% of B-cell lymphomas.CD19 antigen is a well-established target for B-cell lymphomas treatment as well as CD20 antigen.Both CD19-targeting CAR T Cells and CD20-targeting CAR T Cells can be used as adoptive cellular immunotherapies for B-cell lymphomas.Though two kinds of single target treatments were proved can induce recession of B-cell lymphomas, the risk of cancer cells to escape and tumor recurrence are still existed. There are no report about combination transfer of two kinds of single target treatments.This research aimed emphasis on safety and therapeutic efficacy evaluation,as well as if combination transfer can decrease recurrence rate.

DETAILED DESCRIPTION:
To determine:

Primary Outcome Measure:

The Overall complete remission rate and one-year survival rate of combination transfer of CD19-targeting CAR T Cells and CD20-targeting CAR T Cells is superior to or at least not worse than two kinds of single target treatments in the treatment of CD19+/CD20+ B-cell lymphomas.

The risk of cancer recurrence in a year of combination transfer of CD19-targeting CAR T Cells and CD20-targeting CAR T Cells is inferior to two kinds of single target treatments.

Secondary Outcome Measures:

Evaluate the initial effect time, time to disease progression, and life quality improvement of combination transfer compare to single target treatments.

Evaluate the safety and tolerability of combination transfer compare to single target treatments by observation of high fever duration in patients and testing related cell factor level in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 70 Years, Male and female
* Survival time>12 weeks
* B cell lymphomas diagnosed by Physical examination,pathological examination,Laboratory tests and imaging tests
* Chemotherapy failure or recurrent B cell lymphomas
* Creatinine< 2.5mg/dl
* Glutamic-pyruvic transaminase, glutamic oxalacetic transaminase< 3 fold of normal level
* Bilirubin<2.0mg/dl
* Karnofsky Performance Status>50% at the time of screening
* Adequate pulmonary, renal, hepatic, and cardiac function
* Fail in autologous or allogenic haemopoietic stem cell transplantation
* Free of leukocytes removal contraindications
* Voluntarily join CAR-T clinical trial
* Understand and sign written informed consent

Exclusion Criteria:

* Pregnant or nursing women or women with pregnancy plan in half a year
* Any infectious disease (HIV, active tuberculosis, ect.)
* Active hepatitis B, active hepatitis C infection
* Feasibility assessment proves that the efficiency of transduction of lymphocyte is below 10% or the lymphocyte amplification is below 5 fold with the costimulation of cluster of differentiation 3(CD 3)and cluster of differentiation 8(CD 8)
* Abnormal vital signs or cannot cooperate with the inspectors
* mental or psychological disease cannot cooperate with treatment and curative effect evaluation
* Highly allergic constitution or history of severe allergies, especially allergy to interleukin-2(IL-2)
* General infection or local severe infection, or other infection that is not controlled
* Dysfunction in lung, heart, kidney and brain
* Severe autoimmune diseases
* Other symptoms that are not applicable for CAR-T

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall complete remission rate | Half a year
  The complete remission rate will be evaluated by routine methods.

SECONDARY OUTCOMES:
The initial effect time | 1 year
  The initial effect time will be recorded.
The one-year survival rate | 1 year
  The one-year survival rate will be recorded.
The safety and the tolerability(incidence of treatment-emergent adverse events defined as dose-limited toxicity) | 1 month
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
The time to disease progression | 1 year
  The time to disease progression will be counted after complete remission.
The one-year recurrence | 1 year
  The one-year recurrence will be counted after complete remission.
The life quality improvement | 1 year
  The life quality improvement will be evaluated by appetite,sleep,pain and mental state.

CONTACTS AND LOCATIONS:
Overall Officials: Shengqin Ye, M.D., Principal Investigator — Shanghai Longyao Biotechnology Inc., Ltd.
Locations (1):
- Shanghai Longyao Biotechnology Inc., Ltd., Shanghai, Jingan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Zhang WY, Han QW, Liu Y, Dai HR, Guo YL, Bo J, Fan H, Zhang Y, Zhang YJ, Chen MX, Feng KC, Wang QS, Fu XB, Han WD. Effective response and delayed toxicities of refractory advanced diffuse large B-cell lymphoma treated by CD20-directed chimeric antigen receptor-modified T cells. Clin Immunol. 2014 Dec;155(2):160-75. doi: 10.1016/j.clim.2014.10.002. Epub 2014 Oct 16. PMID 25444722
- [Background] Witkowska M, Smolewski P. Emerging immunotherapy and strategies directly targeting B cells for the treatment of diffuse large B-cell lymphoma. Immunotherapy. 2015;7(1):37-46. doi: 10.2217/imt.14.93. PMID 25572478
- [Background] Brudno JN, Somerville RP, Shi V, Rose JJ, Halverson DC, Fowler DH, Gea-Banacloche JC, Pavletic SZ, Hickstein DD, Lu TL, Feldman SA, Iwamoto AT, Kurlander R, Maric I, Goy A, Hansen BG, Wilder JS, Blacklock-Schuver B, Hakim FT, Rosenberg SA, Gress RE, Kochenderfer JN. Allogeneic T Cells That Express an Anti-CD19 Chimeric Antigen Receptor Induce Remissions of B-Cell Malignancies That Progress After Allogeneic Hematopoietic Stem-Cell Transplantation Without Causing Graft-Versus-Host Disease. J Clin Oncol. 2016 Apr 1;34(10):1112-21. doi: 10.1200/JCO.2015.64.5929. Epub 2016 Jan 25. PMID 26811520
- [Background] Hay KA, Turtle CJ. Chimeric Antigen Receptor (CAR) T Cells: Lessons Learned from Targeting of CD19 in B-Cell Malignancies. Drugs. 2017 Mar;77(3):237-245. doi: 10.1007/s40265-017-0690-8. PMID 28110394
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Sang W, Shi M, Yang J, Cao J, Xu L, Yan D, Yao M, Liu H, Li W, Zhang B, Sun K, Song X, Sun C, Jiao J, Qin Y, Sang T, Ma Y, Wu M, Gao X, Cheng H, Yan Z, Li D, Sun H, Zhu F, Wang Y, Zeng L, Li Z, Zheng J, Xu K. Phase II trial of co-administration of CD19- and CD20-targeted chimeric antigen receptor T cells for relapsed and refractory diffuse large B cell lymphoma. Cancer Med. 2020 Aug;9(16):5827-5838. doi: 10.1002/cam4.3259. Epub 2020 Jul 1. PMID 32608579